CLINICAL TRIAL: NCT07146737
Title: Predictive Performance of a Generative Model for Corneal Tomography After Implantable Collamer Lens Implantation
Brief Title: Predictive Performance of a Generative Model for Corneal Tomography After ICL Implantation
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Fu Gui, Associate research fellow; Attending physician, Second Affiliated Hospital of Nanchang University
Other Study IDs: [2025] NO.(86)
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: ICL; Vault; Deep Learning; AI (Artificial Intelligence)
Keywords: Implantable Collamer Lens (ICL) implantation surgery; Corneal tomography; vault; Artificial Intelligence; Deep Learning
MeSH Terms: conditions — T-Lymphocytopenia, Idiopathic CD4-Positive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Eyes with ICL surgeries: Eyes with ICL surgeries which were performed by surgeons with experiences.
  Interventions: Diagnostic Test: Corneal tomography generation model after ICL surgery

INTERVENTIONS:
Diagnostic Test: Corneal tomography generation model after ICL surgery — The ICL procedures collected would be assessed by the corneal tomography generation model. The performance of the model would be assessed, including accuracy,AUC, sensitivity and specificity.

SUMMARY:
To evaluate the efficacy of a corneal tomography Imaging model in predicting postoperative vault based on preoperative corneal topography in Implantable Collamer Lens (ICL) surgery.

DETAILED DESCRIPTION:
Accurate vault prediction is crucial for Implantable Collamer Lens (ICL) surgery safety and efficacy. Current methods using preoperative biometrics and regression formulas show limited accuracy due to parameter variability and incomplete utilization of corneal topography data. To address this, we developed a deep learning model that predicts postoperative vault while generating anterior chamber morphology images from preoperative data, enabling personalized surgical planning.

ELIGIBILITY:
Inclusion Criteria:(1) stable myopia (≤0.50D/year change for 2 years), (2) ACD ≥2.80mm, (3) intact corneal endothelium (≥2000 cells/mm²), and (4) no confounding ocular/systemic conditions.

Exclusion Criteria:(1) glaucoma-spectrum disorders or retinal vasculopathies, (2) prior corneal/intraocular surgery, (3) compromised corneal endothelium, (4) uncontrolled systemic diseases, and (5) pregnancy/lactation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients from clinics in different eye centers across China. Each subject must with complete surgical video recording and medical records.
Sampling Method: Non-Probability Sample
Enrollment: 818 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-07-03 (Actual); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
AUROC of convolutional neural network in predicting vault after ICL surgery | Day 7
  The area under the receiver operating characteristic of convolutional neural network in predicting vault after ICL surgery

SECONDARY OUTCOMES:
Sensitivity and specificity of convolutional neural network in predicting Vault after ICL implantation | Day 7
  Sensitivity and specificity of convolutional neural network in predicting Vault after ICL implantation

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China